CLINICAL TRIAL: NCT00001398
Title: A Phase I/II Trial of Recombinant Methionyl Human Stem Cell Factor (r-metHuSCF) in Patients Diagnosed With Acquired Aplastic Anemia
Brief Title: Stem Cell Factor Medication for Aplastic Anemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 940016; 94-H-0016
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-06

CONDITIONS: Aplastic Anemia; Pancytopenia
Keywords: Hematopoiesis; Stem Cell Cycling; Bone Marrow Failure; Acquired Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic; Pancytopenia; Bone Marrow Failure Disorders | interventions — ancestim

INTERVENTIONS:
Drug: Recombinant Methionyl Human Stem Cell Factor (r-metHuSCF)

SUMMARY:
This trial, sponsored by Amgen, Inc., which produces the recombinant methionyl human stem cell factor (r-metHuSCF), also involves two other institutions. The primary objective is determination of the safety of administering multiple doses of r-metHuSCF in the setting of acquired aplastic anemia and evaluation of the effect of r-metHuSCF on peripheral blood counts. Potential effects of r-metHuSCF on frequency of need for red cell or platelet transfusions and on bone marrow morphology/cellularity will also be evaluated.

DETAILED DESCRIPTION:
This trial, sponsored by Amgen, Inc., which produces the recombinant methionyl human stem cell factor (r-metHuSCF), also involves two other institutions. The primary objective is determination of the safety of administering multiple doses of r-metHuSCF in the setting of acquired aplastic anemia and evaluation of the effect of r-metHuSCF on peripheral blood counts. Potential effects of r-metHuSCF on frequency of need for red cell or platelet transfusions and on bone marrow morphology/cellularity will also be evaluated.

ELIGIBILITY:
Acquired moderate or severe aplastic anemia.

Intolerant to, or failure to durably respond to, ATG/ALG therapy with or without cyclosporin.

Patients may not have received ATG/ALG, therapy for 12 weeks prior to enrollment or cyclosporin for 4 weeks prior to enrollment.

Two years of age or older.

Karnofsky Performance Status greater than or equal to 60 percent.

Adequate organ function as defined by serum creatine less than 2.0 mg/dl and a bilirubin less than 2.0 mg/dl.

Patients (or their parent[s]/responsible guardian[s]) must be able to comprehend and be willing to sign an informed consent prior to starting r-metHuSCF therapy.

No current diagnosis or past history of myelodysplastic syndromes.

No diagnosis of Fanconi's anemia, dyskeratosis congenita, or other congenital forms of aplastic anemia.

No current diagnosis of clinically active paroxysmal nocturnal hemoglobinuria (PNH) defined as patients with clinically significant thrombosis or hemolysis.

No diagnosis of eosinophilic fasciitis.

No treatment with ATG, ALG, or other immunosuppresive agents within 12 weeks of enrollment or treatment with cyclosporine A or IL-3 within 4 weeks of enrollment.

No treatment with hematopoietic growth factors within 2 weeks of enrollment.

No evidence of active uncontrolled infection.

No known allergy to Ecoli-derived products.

No current or recent symptoms of asthma occurring within the past 10 years (including allergic asthma, or asthma induced by cold temperature, infection, or exercise).

No history of anaphylactic/anaphylactoid-type event manifested by disseminated urticaria, laryngeal edema, and/or bronchospasm (or for example: food, insect bites, etc). Patients with drug allergies, manifested solely by rash and/or urticaria, are not excluded. An isolated episode of urticaria occuring more than 3 years earlier is not a contraindication.

No significant nonmalignant disease including previously documented HIV infection, uncontrolled hypertension (diastolic blood pressure greater than 115 mmHg), unstable angina, congestive heart failure (greater than NY Class II), poorly controlled diabetes, coronary angioplasty within 6 months, or uncontrolled atrial or ventricular cardiac arrhythmias.

No pregnancy or breast feeding. Those of childbearing potential must observe adequate birth control measures.

No treatment with an investigational agent (other than hematopoietic growth factors) within 4 weeks of study entry.

No concurrent use of beta adrenergic blocking agents.

No concurrent use, or use within the past 2 weeks, of Monoamine Oxidase Inhibitors (MAO Inhibitors).

No psychiatric, addictive, or any disorder which compromises ability to give truly informed consent for participation in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 1993-10; Study Completion 2002-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Camitta BM, Thomas ED, Nathan DG, Gale RP, Kopecky KJ, Rappeport JM, Santos G, Gordon-Smith EC, Storb R. A prospective study of androgens and bone marrow transplantation for treatment of severe aplastic anemia. Blood. 1979 Mar;53(3):504-14. No abstract available. PMID 32941
- [Background] Camitta BM, Storb R, Thomas ED. Aplastic anemia (first of two parts): pathogenesis, diagnosis, treatment, and prognosis. N Engl J Med. 1982 Mar 18;306(11):645-52. doi: 10.1056/NEJM198203183061105. No abstract available. PMID 7035946
- [Background] Szklo M, Sensenbrenner L, Markowitz J, Weida S, Warm S, Linet M. Incidence of aplastic anemia in metropolitan Baltimore: a population-based study. Blood. 1985 Jul;66(1):115-9. PMID 4005425